CLINICAL TRIAL: NCT05558709
Title: Social-cognitive Functioning: Validation of a New Neuropsychological Test and Prediction of Social Behavioural Disorders in Daily Life
Brief Title: Social-cognitive Functioning: Validation of a New Neuropsychological Test
Acronym: REALSOCOG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP220748
Record Dates: First submitted 2022-09-20; First posted 2022-09-28 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Alzheimer's Disease (AD); Lewy Body Dementia (LBD); Frontotemporal Degeneration (FTD)
Keywords: Neurodegenerative diseases; Social behavior; Social cognition; Neuropsychological assessment
MeSH Terms: conditions — Alzheimer Disease; Lewy Body Disease; Neurodegenerative Diseases; Social Behavior | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients (Experimental): Patients suffering from a neurodegenerative disease (Alzheimer's disease (AD), dementia with Lewy bodies (DCL) or fronto-temporal lobar degeneration (FTD))
  Interventions: Other: REALSOCOG; Other: BCS
- Relatives (Other): Caregivers or relatives of included patients, having regular contact with the patient (≥ 2 times per month).
  Interventions: Other: Hetero-questionnaires

INTERVENTIONS:
Other: REALSOCOG — Patients will be asked to perform the REALSoCog serious game-type social cognition assessment task developed by the LMC2 laboratory (UR 7536). Their performance will be compared to those of control individuals recruited in parallel (independant clinical study: CER-U, IRB N°: 00012020-115). Participants will be asked to think about 16 social situations (6 control situations and 10 experimental situations) encountered in a virtual environment representing a city. REALSoCog can be used on a laptop computer, without any additional technical device.
  Other Names: neuropsychological test
  Arms: Patients
Other: BCS — Social-cognitive tasks from the BCS (Ehrlé et al., 2011) will also be offered to patients to test the concurrent validity of REALSoCog. This battery assesses social cognition. It includes paper-and-pencil tasks.
  Other Names: Social-Cognition Battery
  Arms: Patients
Other: Hetero-questionnaires — Hetero-questionnaires assessing patients' social behavior will be transmitted to their relative or primary caregiver (Godefroy & le GREFEX, 2008; Gury and Ehrlé, in progress of validation) in order to verify the concurrent validity of REALSoCog. These hetero-questionnaires aim to identify and quantify the presence of social skills and behaviour disorders.
  Arms: Relatives

SUMMARY:
It is now established that disturbances in social cognition are frequent in neurology and that they contribute to the development of social conduct disorders. Their assessment is therefore essential, particularly in order to propose early and adapted care. However, this assessment remains limited today. A new serious game-type test, REALSoCog, has been developed to address the shortcomings of current tools and to highlight disturbances in social behaviors. The latter are not always observed in consultation although they are often reported by caregivers. The objective of this research is therefore to validate the REALSoCog task in a pathological population (currently being standardized in the general population: CER-U, IRB N°: 00012020-115). The clinical interest of this task will be tested with a group of patients suffering from a neurodegenerative disease (Alzheimer's disease (AD), dementia with Lewy bodies (DCL), fronto-temporal lobar degeneration (FTD)) in order to assess its sensitivity and specificity in the detection of social-cognitive disturbances, and in particular in terms of social behaviors (detection of social behavioral disorders reported in daily life). The objective is also to document the socio-cognitive profiles in the mentioned diseases thanks to a more ecological test, and to better understand the links between socio-cognitive processes on the one hand, and individual characteristics on the other hand (e.g. mood and social participation).

DETAILED DESCRIPTION:
It is now established that disturbances in social cognition are frequent in neurology and that they contribute to the development of social conduct disorders. Their assessment is therefore essential, particularly in order to propose early and adapted care. However, this assessment remains limited today. A new serious game-type test, REALSoCog, has been developed to address the shortcomings of current tools and to highlight disturbances in social behaviors. The latter are not always observed in consultation although they are often reported by caregivers. The objective of this research is therefore to validate the REALSoCog task in a pathological population (currently being standardized in the general population: CER-U, IRB N°: 00012020-115). The clinical interest of this task will be tested with a group of patients suffering from a neurodegenerative disease (Alzheimer's disease (AD), dementia with Lewy bodies (DCL), fronto-temporal lobar degeneration (FTD)) in order to assess its sensitivity and specificity in the detection of social-cognitive disturbances, and in particular in terms of social behaviors (detection of social behavioral disorders reported in daily life). The objective is also to document the socio-cognitive profiles in the mentioned diseases thanks to a more ecological test, and to better understand the links between socio-cognitive processes on the one hand, and individual characteristics on the other hand (e.g. mood and social participation).

ELIGIBILITY:
Inclusion Criteria:

For patients:

* Patient aged between 18 and 90 years
* Mini Mental State Examination (MMSE) score greater than or equal to 20
* Patient able to express his or her non-opposition to participate in the study in an informed and autonomous manner
* Patient with a neurodegenerative pathology: FTD, AD or LBD.

For caregivers:

* Over 18 years of age
* Regular contact with the patient (≥ 2 times per month)

Exclusion Criteria:

For patients:

* Neurological or psychiatric comorbidity
* Notable sensory disorders (e.g., profound or total deafness, age-related macular degeneration, blindness, etc.) that may interfere with experimental completion.
* Opposition to participation in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-11-28 (Estimated); Primary Completion 2029-11-28 (Estimated); Study Completion 2029-11-28 (Estimated)

PRIMARY OUTCOMES:
rate of inappropriate behavioural intentions | 1 hour and a half
  It is measured by the REALSoCog task through a question asking the participant to specify his behavioral intention in the case where he would have declared his intention to act in front of the social situation presented. These questions are asked for each social situation presented, i.e. for a total of 16 situations

SECONDARY OUTCOMES:
Assessment of Moral cognition | 1 hour and a half
  The ability to detect moral transgressions, the ability to detect conventional transgressions, and the ability to detect control situations (non-transgressive situations) are measured by the question "Does this situation seem appropriate or inappropriate to you?" asked after each REALSoCog situation. The severity judgment of moral transgressions and the severity judgment of conventional transgressions are measured by the question "How inappropriate does it [the situation] seem to you?" asked after each response characterizing the situation presented as inappropriate in REALSoCog.
Evaluation of Empathy and emotional reactivity | 1 hour and a half
  The intensity of emotional empathy and the intensity of emotional reactivity are measured by the question "How much are you affected by the situation? This question is asked after each experimental situation of REALSoCog (i.e. situations involving a transgression and situations constructed to elicit empathy), i.e. for 10 situations.
  The valence and congruence of the emotions felt are measured by the question "The emotion you feel at the sight of this situation is: 1 (very negative) to 5 (very positive)". This question is asked after each experimental situation of REALSoCog (i.e. situations involving a transgression and situations constructed to elicit empathy), i.e. for 10 situations.
Assessment of theory of mind | 1 hour and a half
  The ability to detect the intentionality of an action is measured by the question "Is the behavior of the [main protagonist in the situation] intentional? Yes / No". This question is asked for 5 REALSoCog situations.
  The ability to characterize the valence of this intention and the average valence of the attributed intentions is measured by the question "In your opinion the intention is: 1 (very malicious) to 5 (very benevolent)". This question is asked for 5 REALSoCog situations.
  The ability to infer an affect to others is measured by the question "How does [main protagonist of the situation] feel?". This question is asked for 8 REALSoCog situations.
  The intensity of the affect attributed to others is measured by the question "How does [main protagonist of the situation] feel about [subject's response to the previous question]?" This question is asked for 8 REALSoCog situations.

CONTACTS AND LOCATIONS:
Overall Officials: Marc VERNY, Pr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital de la Pitié-Salpêtrière, Paris, France